CLINICAL TRIAL: NCT05404191
Title: DEVELOPMENT OF A CLINICAL PREDICTION RULES TO IDENTIFY EFFICACY OF LOW LEVEL LASER ON BURN WOUND HEALING
Brief Title: Prediction Rules for Low Level Laser on Burn Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed mohamed nagy, lecturer of physical therapy for surgery- Cairo university, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003532
Record Dates: First submitted 2022-05-03; First posted 2022-06-03 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Burn Wound; Clinical Prediction Rules
MeSH Terms: conditions — Burns | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: 60 adult of both sexes will participate in this study selected from burn unit of AHMED ORABI hospital, Their ages range from 10 to 50 years, TBSA more than 15%, partial thickness burn depth.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- burn wound receiving low level laser therapy (Experimental)
  Interventions: Device: low level laser therapy

INTERVENTIONS:
Device: low level laser therapy — Low level laser therapy will be performed for 30 min 3 times per week for 8 weeks on the wound area.
  Wound area was irradiated by a red 655 nm light, 150 mW, 2 J/cm2 at the bed of the wound.

SUMMARY:
The purpose of this study is to investigate whether patients' age, total burned surface area, wound stage and wound depth determine wound healing response to low level laser therapy in burn patients

DETAILED DESCRIPTION:
It will be hypothesized that

1. Age may significantly affect burn wound healing's response to low level laser therapy.
2. TBSA may significantly affect burn wound healing's response to low level laser therapy.
3. Depth of wound may significantly affect burn wound healing's response to low level laser therapy.
4. Wound healing stage may significantly affect burn wound healing's response to low level laser therapy. There will be only one intervention group. The duration of the study will be 6 weeks divided to 18 sessions (three sessions per week). Sixty patients (male and female) will be recruited from the burn units.

Low level laser therapy will be performed for 30 min 3 times per week for 8 weeks on the wound area.

Wound area was irradiated by a red 655 nm light, 150 mW, 2 J/cm2 at the bed of the wound.

ELIGIBILITY:
Inclusion Criteria:

* Partial thickness Burn wound depth.
* Age ranges from 20-50 years.
* TBSA more than 15%
* Sufficient understanding to perform the test

Exclusion Criteria:

* Diabetic patients.
* Burn wound with skin graft
* Infected wounds
* Patients receiving immunosuppressive drugs.
* Patients receiving irradiation or chemotherapy.
* Chronic circulatory diseases
* Severe associated injury with burn.
* Associated co-morbidities, such as neurological diseases, malnutrition, and other inﬂammatory and/or infectious diseases.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
reduced wound surface area | maximum of 6 weeks
  measure of wound surface area using manual tracing method before and after application of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt